CLINICAL TRIAL: NCT05977127
Title: Intradermal Administration of a COVID-19 mRNA Vaccine in Elderly
Acronym: HVaNa
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment rate dropped because of national COVID-19 vaccination campaign taking place parallel to this study.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-503800-99-00
Record Dates: First submitted 2023-08-03; First posted 2023-08-04 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Vaccination; Infection; COVID-19
Keywords: Intradermal; COVID-19 mRNA vaccine; Elderly; Immune response
MeSH Terms: conditions — Infections; COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Intervention Model Description: open-label, randomised, proof-of-concept intervention study
Masking Description: Only laboratory personnel is masked. Because of the different administration routes it is not possible to mask the participants or investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intradermal vaccination with 20 mcg mRNA vaccine (Experimental): Participants will receive a single dose of 20 mcg COVID-19 mRNA vaccine (Comirnaty; Pfizer/BioNTech) through the intradermal route using microneedles.
  Interventions: Biological: Comirnaty
- Intramuscular vaccination with 30 mcg mRNA vaccine (Active Comparator): Participants will receive a single dose of 30 mcg COVID-19 mRNA vaccine (Comirnaty; Pfizer/BioNTech) through the intramuscular route.
  Interventions: Biological: Comirnaty
- Intramuscular vaccination with 20 mcg mRNA vaccine (Active Comparator): Participants will receive a single dose of 20 mcg COVID-19 mRNA vaccine (Comirnaty; Pfizer/BioNTech) through the intramuscular route.
  Interventions: Biological: Comirnaty

INTERVENTIONS:
Biological: Comirnaty — Administration of Comirnaty vaccine

SUMMARY:
Respiratory tract infections, e.g. caused by SARS-CoV-2, disproportionately affect elderly. Vaccination has shown to be the most cost-effective approach to prevent infections. However, older adults often fail to induce a potent immune response to vaccines, as was also seen recently for COVID-19 mRNA vaccines. This is likely due to immune dysfunction as a consequence of aging. To potentiate a stronger immune response, vaccine administration into the papillary dermis (intradermal, ID) has been proposed as an alternative strategy to intramuscular (IM) administration.

Vaccination through the ID route has shown to be safe and equally or more effective than IM vaccination with a wide variety of vaccines. Recently, ID administration has been tested with two COVID-19 mRNA vaccines (Spikevax, Moderna and Comirnaty, Pfizer/BioNTech) in reduced (fractional) doses of the standard IM dose.

To ease ID administration and thereby facilitate the implementation of this route, silicon-based microneedles have been developed. These needles have shown to allow ID administration of the Spikevax vaccine with equal safety and immunogenicity profiles as the traditional Mantoux approach in young adults.

In the present study, we will investigate the immunogenicity of a 20 mcg dose of the COVID-19 mRNA Comirnaty vaccine through ID administration with silicon microneedles in elderly people (75 years and older), and compare this to immunogenicity of IM administration of a 20 mcg dose and a 30 mcg (standard IM) dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥75 years at the moment of immunization.
* Healthy, determined by medical history and clinical judgement of the investigator. Participants with a pre-existing illness that is stable, defined as disease not requiring significant change in therapy or hospitalisation during the 6 weeks before enrolment and not expected to require any intervention during the study, can be included.
* Willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, and other study procedures.
* Willing to postpone their regular COVID-19 vaccination upon invitation by the Municipal Health Service or general practitioner until at least four months after receiving the intervention.
* Completed a primary series of COVID-19 vaccination.
* Capable and willing to give personal signed informed consent.
* Adequate understanding of the procedures of the study and agrees to abide strictly thereby.
* Fully conversant in the Dutch language.
* Agrees his/her general practitioner is informed about participation in the study.
* Agrees to provide access to information regarding their vaccination background.
* Agrees that the study physician and his/her delegates have access to their medical file at Radboudumc.

Exclusion Criteria:

* Medical or psychiatric condition that may increase the risk of study participation or, in the investigator's judgement, make the participant inappropriate for the study.
* No decision-making capacity.
* History of severe adverse reaction to a vaccine or to any component of the study intervention.
* Thrombose with thrombocytopenia syndrome after vaccination with a COVID-19 vaccine.
* Dermatological conditions that might interfere with the ID vaccination.
* Receipt of COVID-19 vaccination within 3 months before receiving the study intervention.
* Known or suspected immunodeficiency, as determined by medical history or medication use (inhalation corticosteroids are allowed).
* History of autoimmune disease or an active autoimmune disease requiring therapeutic intervention.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate IM injection.
* Participation in other studies involving other study interventions within 28 days prior and during 28 days after receiving the study intervention.
* Receipt of any other non-study vaccine within 28 days prior and after receiving the study intervention.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Concentrations of SARS-CoV-2-Spike protein specific IgG antibodies in serum for the different intervention groups | at 28 days after vaccination

SECONDARY OUTCOMES:
Titers of SARS-CoV-2 specific neutralising antibodies in serum of the different intervention groups | at 28 days after vaccination
The percentage of participants with local and systemic adverse events | up to 28 days after vaccination
  * Solicited adverse events (AEs): local reactions, reaction of regional lymph nodes, and systemic reactions up to 14 days following vaccination
  * Unsolicited AEs up to 28 days following vaccination
  * Serious AEs (SAEs) up to 28 days following vaccination
  * Use of antipyretics and analgesics up to 14 days following vaccination

OTHER OUTCOMES:
Concentrations of SARS-CoV-2-Spike protein specific antibodies in serum and mucosal samples for the different intervention groups at various timepoints | Day 0, day 28 and month 4 after vaccination
Titers of SARS-CoV-2 specific neutralising antibodies in serum and mucosal samples of the different intervention groups at various timepoints | Day 0, day 28 and month 4 after vaccination
Changes in expression level of host genes | day 0 and day 1 after vaccination
Cellular responses in blood and mucosal samples at various timepoints | Day 0, Day 28, month 4 after vaccination
  e.g. expressed as percentages of immune cell subsets or concentration of cytokines
Functional and phenotypic characterization of T cells at various timepoints after vaccination | Day 0, Day 28, month 4 after vaccination
  e.g. expressed as percentages of immune cell subsets or concentration of cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Hans de Graaf, Principal Investigator — Stichting Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided